CLINICAL TRIAL: NCT01952444
Title: An Open-Label, Randomized, Parallel Group Study to Assess the Safety, Tolerability and Pharmacokinetics of ETI-204 Alone and in the Presence of Ciprofloxacin in Adult Volunteers
Brief Title: Safety, Tolerability and PK of Intravenous (IV) ETI-204 Alone and in Presence of Ciprofloxacin in Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Elusys Therapeutics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AH110
Record Dates: First submitted 2013-09-20; First posted 2013-09-30 (Estimated); Results first posted 2019-04-08 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-01

CONDITIONS: Inhalational Anthrax
Keywords: monoclonal antibody, ETI-204, ciprofloxacin, safety, PK
MeSH Terms: conditions — Inhalation anthrax | interventions — obiltoxaximab; Ciprofloxacin

ARMS (2):
- Group 1 ETI-204 and Ciprofloxacin (Experimental): Participants will receive a single IV dose of 16 mg/kg ETI-204 infused over 90 minutes on Day 1, immediately followed by an IV dose of ciprofloxacin 400 mg infused over 60 minutes, followed by oral doses of ciprofloxacin (750 mg every 12 hours) from Day 2 to Day 8 and a final dose on the morning of Day 9.
  Interventions: Biological: ETI-204; Drug: Ciprofloxacin
- Group 2 ETI-204 Alone (Other): Participants will receive a single IV dose of 16 mg/kg ETI-204 infused over 90 minutes on Day 1.
  Interventions: Biological: ETI-204

INTERVENTIONS:
Biological: ETI-204 — A single IV infusion of 16 mg/kg ETI-204 over 90 minutes on Day 1
  Other Names: Obiltoxaximab
Drug: Ciprofloxacin — A single IV Infusion of 400 mg Ciprofloxacin over 60 minutes immediately following the infusion of ETI-204 on Day 1, followed by oral Ciprofloxacin (750 mg every 12 hours) on Days 2-8, and a final oral dose on the morning of Day 9.
  Arms: Group 1 ETI-204 and Ciprofloxacin

SUMMARY:
Evaluate the safety, tolerability and pharmacokinetics (PK) of intravenous (IV) ETI-204 alone and in the presence of IV and oral ciprofloxacin

DETAILED DESCRIPTION:
An open-label, randomized, parallel group study of IV ETI-204 administered alone and in the presence of IV and oral ciprofloxacin in 40 adult volunteers.

Subjects will be randomized to two groups of 20 subjects each in a 1:1 ratio. Group 1 will receive a single IV dose of ETI-204 16 mg/kg followed immediately at the end of the infusion by a single dose of IV ciprofloxacin (400 mg), followed by oral ciprofloxacin (750 mg) every 12 hours on Days 2-8 with the final oral dose on the morning of Day 9. Group 2 will receive IV ETI-204 (16 mg/kg) only.

The total duration of the study for each subject will be approximately 100 days divided as follows:Screening: Days -28 to -2; In-Unit Phases: Days -1, 1 and 2 [all subjects]; Days 8, 9 and 10 [Group 1 only]; Out-of-Unit Visits: Day 9 [Group 2 only]; Day 16 (+/- 3 days); Day 29 (+/- 3 days); Day 43 (+/- 3 days); Final Visit: Day 71 (+/- 3 days).

Following completion of a Screening visit subjects will arrive at the clinical research unit (CRU) on Day -1 following at least a 10-hour fast. On Day 1, subjects who qualify for entry into the study will be randomized to receive either ETI-204 plus IV and oral ciprofloxacin (Group 1) or ETI-204 only (Group 2) in a 1:1 ratio according to the randomization treatment assignment.

On Day 1, all subjects will receive 50 mg oral diphenhydramine approximately 30 minutes prior to ETI-204 infusion. Subjects in Group 1 will receive IV ETI-204 16 mg/kg infused over 90 minutes, immediately followed by IV ciprofloxacin 400 mg infused over 60 minutes. Subjects in Group 2 will receive IV ETI-204 16 mg/kg infused over 90 minutes.

All subjects will be discharged from the CRU on Day 2.

On Days 2 through 8, subjects in Group 1 will receive oral ciprofloxacin (750 mg every 12 hours); the final dose will be received on the morning of Day 9. Oral ciprofloxacin dosing begins 24 hours after the initiation of the ciprofloxacin infusion on Day 1. Subjects in Group 1 will return to the CRU on Day 8 and will be discharged from the unit following completion of PK sampling on Day 10.

Subjects in Group 2 will return to the unit for an out-patient visit on Day 9 but will not be re-admitted to the CRU for an overnight stay.

All subjects will return to the CRU for out-patient visits on Days 16, 29, 43, and 71.

ELIGIBILITY:
Inclusion Criteria:

1. Females or males between 18 and 60 years of age
2. All females, regardless of childbearing potential, must have a negative serum beta human chorionic gonadotropin (β-hCG) pregnancy test at Screening and Day -1
3. Females of childbearing potential (i.e., not postmenopausal or surgically sterile) must agree to practice abstinence or to use a medically accepted method of contraception from the time of Screening through 30 days after the final study visit. Acceptable methods of contraception include diaphragm with spermicide; sponge with spermicide; condom with spermicide; or intrauterine device with condom or spermicide. The following contraceptive methods are acceptable only when used with a condom and spermicide: birth control pills, birth control patches, vaginal ring, hormone under the skin, or hormone injections
4. Postmenopausal females, defined as females who have had amenorrhea for at least 12 months either naturally or following cessation of all exogenous hormonal treatments, and have a follicle-stimulating hormone (FSH) level of > 40 mIU/mL at Screening
5. Females who have undergone surgical sterilization, including hysterectomy, bilateral oophorectomy, bilateral salpingectomy, tubal ligation, or tubal essure ≥ 3 months prior to Screening. Tubal essure requires radiological confirmation of occlusion of the fallopian tubes. Subjects who cannot provide documentation may participate if they agree to follow the methods of contraception specified in Inclusion Criterion #3
6. Males must agree to practice abstinence or use a condom with spermicide and refrain from sperm donation during the study and for 30 days after the final study visit. Note this does not apply to males who have undergone a vasectomy and can provide documentation of confirmatory sperm count 3 months post procedure.
7. Provide written informed consent
8. Willing to comply with study restrictions (see Section 4.5.3 for a complete list of study restrictions)

Exclusion Criteria:

1. Pregnant or lactating woman
2. Clinically-significant comorbidity that would interfere with completion of the study procedures or objectives or compromise the subject's safety
3. Supine systolic blood pressure (BP) ≥ 150 mmHg or ≤ 90 mmHg or diastolic BP ≥ 95 mmHg
4. Use of H1 receptor antagonists (i.e. antihistamines) within 5 days prior to Day 1
5. Evidence of drug or alcohol abuse as determined by the Investigator, within 6 months of Day 1
6. Positive test result for drugs of abuse (with the exception of medically prescribed drugs) at Screening or on Day -1
7. Positive test for alcohol at Screening or Day -1
8. Treatment with an investigational agent within 30 days or five half-lives of the investigational agent at Day 1 (whichever is longer)-
9. Congenital or acquired immunodeficiency syndrome
10. Prior solid organ or bone marrow transplant
11. Positive test for Hepatitis B (surface antigen), Hepatitis C, or human immunodeficiency virus (HIV) at Screening
12. History of prior treatment for anthrax exposure or prior anthrax infection
13. Prior immunization with any approved or investigational anthrax vaccine or prior treatment with an investigational anthrax treatment (i.e., ETI-204, raxibacumab, or anthrax immune globulin)
14. Military personnel deployed in 1990 or after, unless the subject can provide documentation demonstrating they have not previously received any approved or investigational anthrax vaccine
15. Therapeutic use of systemic steroids, immunosuppressive agents, anticoagulants, or anti-arrhythmics within 1 year prior to Day 1; a single short course (i.e., less than 14 days) of systemic steroid therapy is allowed provided it concluded more than 6 months prior to Day 1
16. Donation or loss of > 500 mL of blood within 30 days or plasma within 7 days of Day 1
17. Prior stroke, epilepsy, relapsing or degenerative CNS disease, or relapsing or degenerative ocular disease
18. Myocardial infarction or acute coronary syndrome in the past 5 years, active angina pectoris, or heart failure (New York Heart Association scale > I)
19. History of chronic liver disease
20. Calculated creatinine clearance (CrCl) of < 30 mL/min using the Cockcroft-Gault equation (see Section 5.1)
21. Any clinically significant abnormality, in the Investigator's opinion, on electrocardiogram (ECG) or clinical laboratory tests (hematology, clinical chemistry, or urinalysis) at Screening; out of range results may be repeated to confirm
22. History of allergic or hypersensitivity reactions to other therapeutic antibodies or immunoglobulins
23. History of any malignant neoplasm within the last 5 years, with the exception of adequately treated localized or in situ non-melanoma carcinoma of the skin (e.g. basal cell carcinoma) or the cervix
24. Subjects who, in the opinion of the Investigator, are not suitable candidates for enrollment or who may not comply with the requirements of the study

Exclusion Criteria Specific to the Use of Ciprofloxacin

1. Hypersensitivity to any fluoroquinolone
2. At increased risk of Clostridium. difficile (C. difficile) infection (e.g., prior systemic antibiotic therapy or in-hospital stay of greater than 2 nights over the past 6 months, abdominal surgery within 3 months prior to Day 1, a chronic inflammatory bowel disease or prior C. difficile infection)
3. Any medical condition that may require repeat courses of antibiotics, e.g., recurrent urinary tract or respiratory infections. A short course (i.e.≤ 10 days) of antibiotics within 6 months prior to Day 1 is not exclusionary.
4. A history of any tendon rupture
5. Subjects who smoke or have used tobacco or nicotine containing products within 3 months of Day 1.
6. Use of cation-containing drugs or food supplements within 2 days prior to Day 1
7. Use of protheophylline, theophylline, methylxanthine, tizanidine, or other drugs metabolized via cytochrome P450 1A (CYP1A) within 30 days prior to Day 1
8. Use of glyburide, cyclosporine, didanosine, methotrexate, or probenecid and medications that prolong the QT interval within 30 days prior to Day 1 or within 5 half-lives of Day 1, whichever is longer
9. Subjects at high risk for QT prolongation, including:

   1. Baseline prolongation of QTcF ≥ 500 msec
   2. Risk factors for Torsade de Pointes, including hypocalcemia, hypokalemia, sudden death of unknown cause in a close family member (i.e. biological mother, father or siblings), a near drowning episode, a family history of either Romano-Ward syndrome or Jervell and Lange-Nielson syndrome
   3. The use of concomitant medications that prolong the QT interval within 30 days prior to Day 1

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2013-10-29 (Actual); Primary Completion 2014-04-09 (Actual); Study Completion 2014-04-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Mathews, MD, Principal Investigator — Quintiles, Inc.; Jolene Berg, MD, Principal Investigator — Davita Clinical Research
Locations (1):
- Quintiles, Overland Park, Kansas, United States

REFERENCES:
- [Derived] Nagy CF, Leach TS, Hoffman JH, Czech A, Carpenter SE, Guttendorf R. Pharmacokinetics and Tolerability of Obiltoxaximab: A Report of 5 Healthy Volunteer Studies. Clin Ther. 2016 Sep;38(9):2083-2097.e7. doi: 10.1016/j.clinthera.2016.07.170. Epub 2016 Aug 24. PMID 27568215

RESULTS

PARTICIPANT FLOW:
Groups:
- ETI-204: IV infusion of 16 mg/kg ETI-204
  IV Ciprofloxacin: IV Infusion of 400 mg ciprofloxacin
  Oral Ciprofloxacin: Oral ciprofloxacin (750 mg) every 12 hours on Days 2-8 and final dose on morning of Day 9
- ETI-204 and Ciprofloxacin: IV infusion of 16 mg/kg ETI-204 followed by IV infusion of ciprofloxacin followed by oral ciprofloxacin
  ETI-204: IV infusion of 16 mg/kg ETI-204
Period: Overall Study
Arm/Group | ETI-204 | ETI-204 and Ciprofloxacin
Started | 20 | 20
Completed | 20 | 19
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- ETI-204: Participants received 16 mg/kg ETI-2041 by IV infusion over 90 minutes
- ETI-204 + Ciprofloxacin: Participants received 16 mg/kg ETI-204 by IV infusion over 90 minutes followed by IV infusion of 400 mg ciprofloxacin followed by oral ciprofloxacin (750 mg) every 12 hours on Days 2-8 and a final dose on the morning of Day 9
- Total: Total of all reporting groups
Arm/Group | ETI-204 | ETI-204 + Ciprofloxacin | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 33 (11.8) | 33 (14.0) | 33 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 12 | 12 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 6 | 7
  Not Hispanic or Latino | 19 | 14 | 33
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 3 | 4
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 3 | 8
  White | 14 | 14 | 28
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40
Body Weight [Mean (Standard Deviation); unit: kg] | 78.4 (16.63) | 75.8 (18.26) | 77.1 (17.29)
Height [Mean (Standard Deviation); unit: cm] | 169.5 (7.29) | 169.4 (9.11) | 169.4 (8.15)
BMI [Mean (Standard Deviation); unit: kg/m2] | 27.1 (4.80) | 26.2 (4.75) | 26.7 (4.74)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Adverse Events
Description: Safety was assessed for all subjects in the Safety Population by collecting and monitoring vital signs, clinical laboratory tests, ECGs, physical assessments, skin assessments, infusion site assessments, and adverse events (AEs).
Time Frame: Up to 71 days or 101 days (30 days after the final study visit) for subjects with ongoing adverse events at the final study visit, for each group.
Population: All randomized subjects who received study drug were included in the Safety Population.
Measure: Count of Participants; unit: Participants
Groups:
- ETI-204 + Ciprofloxacin: Participants received 16 mg/kg ETI-204 by IV infusion over 90 minutes followed by IV infusion of 400 mg ciprofloxacin followed by oral ciprofloxacin (750 mg) every 12 hours on Days 2-8 and a final dose on the morning of Day 9. All participants received 50 mg oral diphenhydramine as a required premedication before ETI-204 infusion.
- ETI-204: Participants received 16 mg/kg ETI-204 by IV infusion over 90 minutes. All participants received 50 mg oral diphenhydramine as a required premedication before ETI-204 infusion.
Arm/Group | ETI-204 + Ciprofloxacin | ETI-204
Number analyzed (Participants) | 20 | 20
Participants | 14 | 13

2. Secondary Outcome: Maximum Observed Plasma Concentration of ETI-204 (Cmax)
Description: Blood samples were obtained and serum concentrations were determined using a validated enzyme-linked immunosorbent assay method with an assay range of 100 ng/mL to 5000 ng/mL.
Time Frame: On Day 1 at predose, at the end of ETI-204 infusion, 2.5, 4.5 and 7.5 hours after the start of the ETI-204 infusion, and on Days 2 (24 hours), 9, 16, 29, 43, and 71.
Population: The Pharmacokinetic (PK) Population consisted of all subjects who received ETI-204 and had at least one valid PK parameter. Two subjects in the ETI-204 + ciprofloxacin group received partial doses of ETI-204 (discontinued study drug due to AEs) and were excluded from the PK Population.
Measure: Mean (Standard Deviation); unit: µg/mL
Groups:
- ETI-204 Alone: Participants received 16 mg/kg ETI-2041 by IV infusion over 90 minutes.
Arm/Group | ETI-204 + Ciprofloxacin | ETI-204 Alone
Number analyzed (Participants) | 18 | 20
µg/mL | 397 (63.7) | 402 (91.0)

3. Secondary Outcome: Time to Maximum Observed Plasma Concentration of ETI-204 (Tmax)
Description: as for outcome 2
Time Frame: as for outcome 2
Population: The PK Population consisted of all subjects who received ETI-204 and had at least one valid PK parameter. Two subjects in the ETI-204 + ciprofloxacin group received partial doses of ETI-204 (discontinued study drug due to AEs) and were excluded from the PK Population.
Measure: Median (Full Range); unit: days
Arm/Group | ETI-204 + Ciprofloxacin | ETI-204 Alone
Number analyzed (Participants) | 18 | 20
days | 0.104 [0.0625 to 1.00] | 0.104 [0.0625 to 1.00]

4. Secondary Outcome: Area Under the Concentration-Time Curve From Time 0 to Time of Last Measurable Concentration (AUC0-last))
Description: as for outcome 2
Time Frame: as for outcome 2
Population: All subjects who received ETI-204 and had at least one valid PK parameter were included in the PK Population: Two subjects who received a partial dose of ETI-204 due to AEs and 1 who withdrew prematurely on Day 1 for personal reasons after the IV infusions of ETI-204 and ciprofloxacin were excluded from the ETI-204 + ciprofloxacin group.
Measure: Mean (Standard Deviation); unit: µg.day/mL
Arm/Group | ETI-204 + Ciprofloxacin | ETI-204
Number analyzed (Participants) | 17 | 20
µg.day/mL | 4603 (791) | 4514 (792)

5. Secondary Outcome: Area Under the Concentration-Time Curve From Time 0 to Infinity (AUC0-inf)
Description: as for outcome 2
Time Frame: as for outcome 2
Population: All subjects for whom Cmax, Tmax and AUC0-last were calculated minus 2 subjects (1 in the ETI-204 group and 1 in the ETI-204 + ciprofloxacin group) whose t1/2 values were > than 50% of the total sample collection interval. AUC0-inf and AUC0-inf-based parameters were not reported for those subjects in accordance with the statistical analysis plan.
Measure: Mean (Standard Deviation); unit: µg.day/mL
Arm/Group | ETI-204 + Ciprofloxacin | ETI-204 Alone
Number analyzed (Participants) | 16 | 19
µg.day/mL | 4990 (942) | 4891 (897)

6. Secondary Outcome: Terminal Half-life (t1/2)
Description: as for outcome 2
Time Frame: as for outcome 2
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: days
Arm/Group | ETI-204 + Ciprofloxacin | ETI-204 Alone
Number analyzed (Participants) | 16 | 19
days | 19.0 (3.00) | 19.5 (4.14)

7. Secondary Outcome: Systemic Clearance (CL)
Description: as for outcome 2
Time Frame: as for outcome 2
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Liters/day
Arm/Group | ETI-204 + Ciprofloxacin | ETI-204 Alone
Number analyzed (Participants) | 16 | 19
Liters/day | 0.247 (0.0732) | 0.268 (0.0583)

8. Secondary Outcome: Volume of Distribution (Vd)
Description: as for outcome 2
Time Frame: as for outcome 2
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | ETI-204 + Ciprofloxacin | ETI-204 Alone
Number analyzed (Participants) | 16 | 19
Liters | 6.59 (1.34) | 7.57 (2.58)

9. Secondary Outcome: Volume of Distribution at Steady State (Vss)
Description: as for outcome 2
Time Frame: as for outcome 2
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | ETI-204 + Ciprofloxacin | ETI-204 Alone
Number analyzed (Participants) | 16 | 19
Liters | 5.68 (0.986) | 6.28 (1.68)

10. Secondary Outcome: Number of Participants With Anti-ETI-204 Antibodies
Description: Serum anti-ETI-204 antibody titers were determined for all subjects in the Safety Population. Blood samples were collected and serum samples were assayed at an initial dilution of 1:10. Samples that were positive at the 1:10 dilution were serially diluted 1:2 and assayed until a negative result was attained. The titer of the most dilute sample yielding a positive result was recorded as the titer for that time point. Immunogenicity was measured by the number of participants in each study arm with anti-ETI-204 antibody values post-treatment ≥ 4-times higher than baseline at Day 8, 43 or 71, or if the titer was negative at baseline, the post-treatment sample(s) required a titer of at least 1:20 for it to be considered positive.
Time Frame: On Day 1 at predose and on Days 9, 29, 43, and 71.
Population: All subjects who received ETI-204 and were included in the Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | ETI-204 + Ciprofloxacin | ETI-204 Alone
Number analyzed (Participants) | 20 | 20
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: 71 days or up to 101 days (30 days after the final study visit) for adverse events ongoing at the final study visit, for each group.
Arm/Group | ETI-204 + Ciprofloxacin | ETI-204 Alone
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 14/20 | 13/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ETI-204 + Ciprofloxacin (N=20) | ETI-204 Alone (N=20)
Somnolence (Nervous system disorders) | 5 (5) | 6 (6)
Upperrespiratory tract infection (Infections and infestations) | 2 (2) | 5 (6)
Urticaria (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dizziness postural (Nervous system disorders) | 1 (1) | 0 (0)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vaginitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Vessel puncture site bruise (General disorders) | 0 (0) | 1 (1)
Vulvovaginal mycotic infection (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The data generated in this clinical study are the exclusive property of the Sponsor and are confidential. Written approval from the Sponsor is required prior to disclosing any information related to this clinical study.